CLINICAL TRIAL: NCT04862559
Title: A Prospective, Single Center, Non-randomized, Single Arm, Open Label, Study to Evaluate the Safety and Effectiveness of the NovaCross™ Micro-catheter in Facilitating Crossing Chronic Total Occlusion (CTO) Coronary Lesions
Brief Title: A Single Center Study to Evaluate the Safety of the NovaCross Microcatheter in Crossing Chronic Total Occlusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nitiloop Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NT-CLP-02
Record Dates: First submitted 2021-04-23; First posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2016-09

CONDITIONS: Chronic Total Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NovaCross (Experimental): Subjects in this arm are treated with the investigational device, NovaCross micro-cetheter, to facilitate the opening of a chronic total occlusion (CTO)
  Interventions: Device: NovaCross

INTERVENTIONS:
Device: NovaCross — A device that is intended to asisst interventional cardiologists during catheterization to cross and open coronary chronic total occlusions

SUMMARY:
This is an open label, single-center, prospective, pivotal study in which the investigational device, NovaCross™ micro-catheter, will be tested in up to 15 patients scheduled to undergo CTO-PCI using an anterograde approach.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 25-80
* Patient understands and has signed the study informed consent form.
* Patient is a suitable candidate for non-emergent, coronary angioplasty
* Patient has an angiographic documented Chronic Total Occlusion (i.e. >3 months occlusion duration either by documentation or PI assessment Investigator) showing distal TIMI flow 0.
* Coronary angiography of CTO lesion reveals satisfactory distal vessel visualization
* CTO lesion is located in a coronary vessel with a reference diameter of at least 2 millimeters.
* CTO lesion is suitable for antegrade approach.
* Left ventricle ejection fraction > 25%
* Body Mass Index (BMI) < 40

Exclusion Criteria:

* Patient unable to give informed consent.
* Patient is participating in another study with any investigational drug or device.
* Patient is known or suspected not to tolerate the contrast agent.
* Aorto-ostial CTO location (Ostial bifurcation origins may be considered), SVG CTO.
* Intolerance to Aspirin and/or inability to tolerate a second antiplatelet agent (Clopidogrel and Prasugrel and Ticagrelor).
* Appearance of a fresh thrombus or intraluminal filling defects.
* Recent major cerebrovascular event (stroke or TIA within 30 days)
* Significant anemia (hemoglobin < 8.0 mg / dl)
* Unstable angina requiring emergent percutaneous trans-luminal coronary angioplasty (PTCA) or coronary artery bypass graft (CABG)
* Recent myocardial infarction (MI) (within the past two weeks)
* Unwillingness or inability to comply with any protocol requirements
* Pregnancy or nursing

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2017-09-17 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Adverse Events (Primary Safety) | 30 days
  Accumulative incidence of Major Adverse Cardiovascular Events (MACE), defined as the composite of death, myocardial infarction (MI), or urgent revascularization (target vessel revascularization (TVR) or urgent coronary artery bypass surgery (CABG)).
Technical Success (Primary Efficacy) | 1 day
  Intra-procedural technical success, defined as the ability of the NovaCross™ microcatheter to successfully facilitate placement of a guidewire beyond a native coronary chronic total occlusion in the true vessel lumen

SECONDARY OUTCOMES:
Procedural Success | 1 day
  The ability to cross the lesion with a guidewire in the true lumen, effectively dilate the CTO lesion, and place a coronary stent with residual lumen stenosis of less than 30% while restoring antegrade TIMI 3 flow
Assistance in Guidewire Penetration | 1 day
  The ability of the NovaCross™ micro-catheter to facilitate a guidewire successfully penetrating the proximal cap of the CTO
Crossability | 1 day
  The effectiveness of the extendable portion in intra-CTO microcatheter crossability
Procedual Visualization | 1 day
  The ability to have full visualization of the NovaCross during the CTO procedure
Operator Ease of Use | 1 day
  Assess the usability of the NovaCross™ by the operator
Device Related Perforation Rate | 1 day
  Device-related perforation at the site of target coronary lesion and/or its proximal reference segment

CONTACTS AND LOCATIONS:
Overall Officials: Chanan Schneider, Mr., Study Director — Company Employee
Locations (1):
- Szpital Uniwersytecki w Krakowie, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No